CLINICAL TRIAL: NCT04150484
Title: Influence of an Intervention on Diet, Physical Exercise and Mindfulness in the Quality of Life of Survivors With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Julia Ruiz Vozmediano, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 040907
Record Dates: First submitted 2019-10-20; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Nutrition Related Cancer; Physical Activity; Mindfulness
Keywords: breast cancer survival; mediterranean diet; physical activity; mindfulness
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Diet, Mediterranean; Exercise

STUDY DESIGN:
Intervention Model Description: Patients between 18 and 70 years of age with breast cancer II-III operable in follow-up, seen in the Oncology service of the Virgen de las Nieves Hospital in Granada and residents in the city or metropolitan area of Granada, which had completed, in the 12 months prior to its inclusion, treatment with surgery, radiotherapy and / or systemic chemotherapy treatment (including biological treatment).
  Randomized assignment was made based on age, stage, hormone receptor and her2 status, establishing two groups: a group of dietary intervention, physical exercise and mindfulness and another control group. A longitudinal follow-up was carried out for 6 months from the beginning of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Other): dietary intervention, physical exercise and mindfulness
  Interventions: Other: Mediterranean diet, physical exercise and mindfulness workshops
- control group (No Intervention): Group without any intervention.

INTERVENTIONS:
Other: Mediterranean diet, physical exercise and mindfulness workshops — a group of dietary intervention, physical exercise and mindfulness and another control group, and a longitudinal follow-up was carried out for 6 months from the beginning of the intervention.
  Arms: interventional group

SUMMARY:
ABSTRACT

BACKGROUND:

Breast Cancer (BC) is one of the leading causes of death among women around the world. Integrative oncology, together with conventional medical treatment, has proven to be an important support for the control of cancer symptoms, improvement of quality of life, and contribution to the overall patient health, providing an integrated patient care both physically and emotionally.

METHODS:

75 stage II-III breast cancer survivors were randomized (according to age, tumor stage and receptor status) into 2 groups: intervention and control. Within the intervention group (IG) a diet, exercise and mindfulness intervention was performed, while the control group (CG) did not receive any sort of treatment, during 6 months. Passed (at the beginning and end of the research) questionnaires concerning general health, quality of life (EORTC QLQ-C30 and BR23), and diet (Mediterranean diet adherence test and 24-h-recall) and a blood and urine sample was collected to analyze general biochemical variables.

RESULTS:

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age
* Breast cancer IIA-IIB operable in follow-up
* Seen in the Oncology service of the Virgen de las Nieves Hospital in Granada
* Residents in the city or metropolitan area of Granada
* Had completed, in the 12 months prior to its inclusion, treatment with surgery, radiotherapy and / or systemic chemotherapy treatment (including biological treatment).

Exclusion Criteria:

* Those who presented some physical or psychic limitation that prevented the intervention from being carried out were excluded from the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
Quality of life test (EORTC QOL-C30) | 6 months
  It includes 30 items that are grouped into five scales functional (physical, social, emotional functioning, cognitive and role), three scales of symptoms (fatigue, pain, nausea and vomiting), a global scale of health / quality of life and a number of related individual items with the symptoms of the disease and its treatment, as well as an item of economic impact. The answers to the items on the scales refer to "last week," except the patient's physical functioning scale whose time frame is the present. These answers they obey a Likert format, which ranges from 1 ("Not at all") and 4 ("A lot")

SECONDARY OUTCOMES:
Mediterranean diet adherence test | 6 months
  Adherence to the traditional Mediterranean diet was assessed by a 14-point Mediterranean-diet scale that incorporated the salient characteristics of this diet (range of scores, 0 to 1, with higher scores indicating greater adherence)
Levels of glucose | 6 months
  Levels of glucose mg/dl
Levels of triglycerides | 6 months
  Levels of triglycerides mg/dl
Levels of cholesterol | 6 months
  Levels of cholesterol mg/dl
24 hours recall | 6 months
  Retrospective and quantitative recording method of food and beverage consumption. It consists of remembering all the foods and drinks that were taken the day before.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Ruiz Vozmediano, Dr, Principal Investigator — Hospital Virgen de las Nieves

IPD SHARING:
Plan to Share IPD: Yes
All IPD that and underlie result in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Depends of the journal
Access Criteria: Depends of the journal

REFERENCES:
- [Derived] Ruiz-Vozmediano J, Lohnchen S, Jurado L, Recio R, Rodriguez-Carrillo A, Lopez M, Mustieles V, Exposito M, Arroyo-Morales M, Fernandez MF. Influence of a Multidisciplinary Program of Diet, Exercise, and Mindfulness on the Quality of Life of Stage IIA-IIB Breast Cancer Survivors. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420924757. doi: 10.1177/1534735420924757. PMID 32462950